CLINICAL TRIAL: NCT04346823
Title: Effect of Sevoflurane on the Success of External Cephalic Version for Breech Presentation
Brief Title: Sevoflurane and Success of External Cephalic Version (ECV)
Acronym: ECV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Adel Alqarni, Assistant professor and consultant of anesthesia, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sevoflurane for ECV
Record Dates: First submitted 2020-02-26; First posted 2020-04-15 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Version of Uterus
Keywords: Sevoflurane
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane (Experimental): Each participant started by preoxygenation of 100% oxygen for 3 minutes. Then, parturients breath 1% of sevoflurane in mixture of oxygen and air (FIO2 0.5) by tight face mask with a gas flow of 6 L/min. Values of inspired (FI) and end-tidal (FET) concentrations of sevoflurane, oxygen and respiratory rate (RR) measured by end-tidal carbon dioxide (EtC02) were monitored continuously and recorded at 30 seconds intervals by a gas analyzer.
  30 seconds after stating inhalation sedation, the obstetrician will be asked to start the procedure. HR, FI and FET concentration of sevoflurane, Sp02 and EtC02 will be recorded at 30-s interval during ECV. Non-invasive BP will be recorded every one minute. Duration of ECV in addition to level of difficulty estimated by obstetrician will be recorded.
  ECV considered successful when a cephalic presentation, confirmed by ultrasound scan, achieved.
  Interventions: Drug: Sevoflurane
- No sevoflurane (No Intervention): If the parturient is assigned to the control (nonintervention) group, the participants will not receive any medications neither tocolytics nor analgesics as the routine care in our hospital. However, the participants will be monitored throughout the procedure for vital signs and for pain scores as in the intervention group.

INTERVENTIONS:
Drug: Sevoflurane — Each participant started by preoxygenation of 100% oxygen for 3minutes. Then, parturients breath 1% of sevoflurane in a mixture of oxygen and air (FIO2 0.5) by tight face mask with a gas flow of 6 L/min.
  Thirty seconds after stating inhalation sedation, the obstetrician will be asked to start the procedure.The duration of ECV in addition to the level of difficulty estimated by obstetricians will be recorded. Usually, the duration of ECV does not exceed 10 minutes.
  The intervention will be stopped if the woman reported severe pain, if version could not be achieved readily, or if prolonged fetal bradycardia, uterine bleeding or placental abruption occurred.
  Parturient will be kept in Post Anesthesia Care Unit (PACU) for 45minutes. CTG will be monitored during PACU stay.
  Other Names: Sevorane
  Arms: Sevoflurane

SUMMARY:
External cephalic version (ECV) is noninvasive procedure aiming to turn the fetus to cephalic presentation, thereby enabling vaginal delivery and avoiding unnecessary cesarean delivery. The American College of Obstetricians and Gynecologists (ACOG) suggested that all women near term with breech presentation should be offered a version (9). Its success rate depends on the experience of obstetrician in addition to maternal factors. Several interventions have been tried to increase the success rate of ECV, including but not limited to tocolytics and neuraxial anesthesia. Although parenteral β stimulants and spinal anesthesia proved to be effective for increasing the success rate ECV, their success rates are still not high (10, 11) Sevoflurane's pleasant odor, lack of pungency, and potent bronchodilating characteristics make sevoflurane administration via the facemask for either sedation or induction of anesthesia is suitable. Sevoflurane has sedative and uterine relaxation effects all together would facilitate ECV and consequently would increase its success rate. To the best our knowledge sevoflurane has never been studied for ECV. Up to 1% concentration of sevoflurane has been used for labor analgesia without excessive sedation (8). Therefore, the investigators aim at comparing the success rate of ECV at 36-40 weeks of gestation under 1% of sevoflurane with a control group (received no anesthetic or other obstetric interventions). Other outcomes such as pain score and maternal and fetal complications will also be evaluated.

DETAILED DESCRIPTION:
Pre- procedure all parturients will be asked to be fasting for 8 hours for solid and 2 hours for clear liquids. Before ECV (as routinely done in ECV procedure), a cardiotocogram (CTG) and obstetric ultrasound will be done to confirm the fetal wellbeing and fetal position prior to procedure. The mother and fetus were monitored for at least 30 min before attempting ECV. The procedure will be performed by one of two experienced obstetricians. Fetal heart rate will be recorded throughout the procedure.

In the operating room, standard monitoring will be placed, as well as intravenous line will be established on an upper limb. Baseline measures of BP, HR, O2 Saturation will be taken before proceeding to inhalation sedation, including 3 baseline blood pressure readings to determine baseline values. A circle system, including antibacterial filter and scavenging system is connected to the anesthesia machine (Datex-Ohmeda).

If the parturient is assigned to the control (nonintervention) group, the participants will not receive any medications neither tocolytics nor analgesics as we do routinely in our hospital. However, these participants will be monitored throughout the procedure for vital signs and for pains scores as in the intervention group (see below).

In the intervention group, each participant started by preoxygenation of 100% oxygen for 3minutes. Then, parturients breath 1% of sevoflurane in mixture of oxygen and air (FIO2 0.5) by tight face mask with a gas flow of 6 L/min. Values of inspired (FI) and end-tidal (FET) concentrations of sevoflurane, oxygen and respiratory rate (RR) measured by end-tidal carbon dioxide (EtC02) were monitored continuously and recorded at 30 seconds intervals by a gas analyzer.

Thirty seconds after stating inhalation sedation, the obstetrician will be asked to start the procedure. HR, FI and FET concentration of sevoflurane, Sp02 and EtC02 will be recorded at 30 seconds intervals during ECV. Non-invasive BP will be recorded every one minute. The duration of ECV in addition to the level of difficulty estimated by obstetrician will be recorded. In noninterventional (control) group, the patients will not receive any medication or anesthetic intervention however their vital signs including Sp02, BP and HR will be monitored throughout the procedure at the same interval used for the intervention group, their pain score will be measured as in the intervention group (see below).

A hypotensive episode will be defined as 2 consecutive systolic BP (SBP) measurements less than 20% below the baseline value. The treatment of hypotension consists of Phenylephrine 1 mcg/kg IV bolus will be administered if HR > 60 bpm or Ephedrine 5 mg IV bolus if HR is < 60 bpm. If only the HR is < 55 bpm, but SBP is normal, Glycopyrrolate 0.2 mg IV bolus will be administered.

ECV considered successful when a cephalic presentation, confirmed by ultrasound scan, achieved. Pain intensity measured by VAS will be recorded at the end of procedure and 10 minutes after. In addition, the women's level of satisfaction with the procedure will be assessed using another numerical rating scale (0 = completely dissatisfied, 10 = completely satisfied) 10 min after the end of attempted ECV.

The intervention will be stopped if the woman reported severe pain, if the version could not be achieved readily, or if prolonged fetal bradycardia, uterine bleeding or placental abruption occurred.

Parturient will be kept in the Post Anesthesia Care Unit (PACU) for 45minutes. CTG will be monitored during PACU stay. Maternal oxygen saturation will be measured continuously using pulse oximetry, episodes of hypoxia (Sp02 ≤95%) and need for oxygen therapy will be recorded. Blood pressure will be measured every 5 min; hypotension was defined as a fall in blood pressure of >20% from baseline and will be treated as perioperative period (see above). Isolated bradycardia with HR < 50 bpm will be treated by glycopyrrolate 0.2mg IV bolus. Nausea and vomiting will be documented as adverse effects, regardless of when they occurred, and were treated with intravenous ondansetron 4 mg. Other maternal side effects including drowsiness and dizziness were also documented.

Data Collection Pre-procedure and intra-procedure and post-procedure data will be collected by an anesthesia resident, or an anesthesiologist Not involved in the procedure.

* Pre-procedure data:

  * Age, weight, height, gestation, gravida, parity
  * Estimated fetal weight
  * Number of prior cesarean deliveries
  * Reason for the ECV
* Intra-procedure data:

  * HR, Sp02, EtC02 for RR, FI and FET concentration of sevoflurane will be recorder every 30 seconds
  * BP every one minute
  * Episode of tachycardia
  * Episode of hypotension
  * Episode of desaturation (Sp02 ≤95%)
  * Nausea or vomiting
  * Use of ondansetron
  * Pain intensity measured by VAS
  * Transient fetal bradycardia
  * Emergency Cesarean delivery
* Post-procedure data:

  * HR, RR, Sp02, BP will be recorded every 5 minutes
  * Pain score measured by VAS 10 minutes after ECV
  * Episodes of desaturation
  * Episodes of hypotension
  * Nausea or vomiting
  * Drowsiness
  * Dizziness
  * Fetal bradycardia
  * Maternal satisfaction by using numerical rating scale 0-10 (see above) 10 min after the end of attempted ECV
  * Mode of delivery after successful and failed ECV will be recorded by reviewing the electronic medical records

Randomization:

- Randomization will be achieved by a statistician using an online random number generator

Sample Size Estimation A sample size of 40 parturients (20 per group) would give 80% power to detect a difference of 0.2 in the change in successful ECV rate.

Assuming the use of sevoflurane will have 65% success rate and confidence interval 95% with 5% margin of error and total number of cases per year in our center is 45 patients. The average success rate of ECV in patients who either did not receive any intervention or just receive intravenous analgesia is 43.1% (10). So, we are aiming to increase the success rate of ECV by using Sevoflurane to be more than or equal to 65%.

The sample size calculation will be 40 cases. The sample size was calculated by the help of this website (http://www.raosoft.com/samplesize.html).

Statistical Analysis

This prospective randomized controlled study will compare the difference in success rate of ECV when a subject receives a sevoflurane or not. Other covariable like pain scores and adverse effects will also be recorded. Data will be stored in an excel database and analyzed with SPSS statistical software.

Demographic data and intraoperative and PACU continuous and categorical data will be analyzed by Student t-test, ANOVA for repeated measures, or Chi-Squared test, accordingly.

A P-value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* ASA status I or II (healthy women or patient with mild well-controlled systemic disease)
* Elective ECV
* 36 to 40 weeks of gestation

Exclusion Criteria:

* Multifetal gestation
* Morbid obesity (BMI > 40 at first prenatal medical visit)
* Oligohydramnios or polyhydramnios (AFI <5 cm or > 23 cm)
* Fetal weight >4200g
* Active labor
* Uterine tumors or anomalies
* Abnormal placentation such as Placenta accreta/Previa
* Placental abruption
* Intrauterine fetal death
* Known allergy to sevoflurane
* History of malignant hyperthermia
* Administration of any tocolytics before or during ECV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
The success rate of ECV under sevoflurane compared with that without sevoflurane in parturient undergoing elective ECV at 36-40 weeks of gestation. | 20 minutes
  ECV considered successful when a cephalic presentation assessed by direct palpation of maternal abdominal wall by obstetrician and confirmed by ultrasound scan is achieved.

SECONDARY OUTCOMES:
The pain score (by using visual analogue scale) during ECV under sevoflurane versus that during ECV without sevoflurane | 20 minutes
  The visual analogous scale used for this study measures from 0-10 the intensity of the pain. Where, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10).
The duration of ECV under sevoflurane versus without sevoflurane | 10 minutes
  The duration of ECV procedure in minutes
The maternal satisfaction during ECV procedure between sevoflurane group versus control group | 20 minutes
  The women's level of satisfaction with the procedure will be assessed using numerical rating scale (0 = completely dissatisfied, 10 = completely satisfied)
The incidence rate of complications related to ECV between sevoflurane group versus control group | 45 minutes
  These complications include such as placental abruption, cord prolapse, abnormal cardiotocography, fetomaternal transfers and stillbirth
The incidence of adverse effects after administration of sevoflurane for ECV with that of control group. | 45 minutes
  Possible adverse effects such as nausea, vomiting, drowsiness, hypotension and aspiration pneumonia.
The mode of delivery (vaginal or cesarean) after successful ECV between sevoflurane versus control group | 2 months
  mode of delivery might be either normal vaginal delivery or by cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Adel Alqarni, MD, Principal Investigator — King Saud University

REFERENCES:
- [Background] United States Food and Drug Administration. FDA drug safety communication: FDA review results in new warnings about using general anesthetics and sedation drugs in young children and pregnant women. Updated 2016. Accessed February/10, 2017.
- [Result] Hofmeyr GJ, Kulier R, West HM. External cephalic version for breech presentation at term. Cochrane Database Syst Rev. 2015 Apr 1;2015(4):CD000083. doi: 10.1002/14651858.CD000083.pub3. PMID 25828903
- [Result] Hannah ME, Hannah WJ, Hewson SA, Hodnett ED, Saigal S, Willan AR. Planned caesarean section versus planned vaginal birth for breech presentation at term: a randomised multicentre trial. Term Breech Trial Collaborative Group. Lancet. 2000 Oct 21;356(9239):1375-83. doi: 10.1016/s0140-6736(00)02840-3. PMID 11052579
- [Result] Gregory KD, Jackson S, Korst L, Fridman M. Cesarean versus vaginal delivery: whose risks? Whose benefits? Am J Perinatol. 2012 Jan;29(1):7-18. doi: 10.1055/s-0031-1285829. Epub 2011 Aug 10. PMID 21833896
- [Result] Melo P, Georgiou EX, Hedditch A, Ellaway P, Impey L. External cephalic version at term: a cohort study of 18 years' experience. BJOG. 2019 Mar;126(4):493-499. doi: 10.1111/1471-0528.15475. Epub 2018 Oct 23. PMID 30223309
- [Result] Toscano A, Pancaro C, Giovannoni S, Minelli G, Baldi C, Guerrieri G, Crowhurst JA, Peduto VA. Sevoflurane analgesia in obstetrics: a pilot study. Int J Obstet Anesth. 2003 Apr;12(2):79-82. doi: 10.1016/S0959-289X(02)00195-4. PMID 15321492
- [Result] Suehara T, Morishita J, Ueki M, Ueno M, Maekawa N, Mizobuchi S. Effects of sevoflurane exposure during late pregnancy on brain development of offspring mice. Paediatr Anaesth. 2016 Jan;26(1):52-9. doi: 10.1111/pan.12785. Epub 2015 Oct 13. PMID 26645425
- [Result] Lee S, Chung W, Park H, Park H, Yoon S, Park S, Park J, Heo JY, Ju X, Yoon SH, Kim YH, Ko Y. Single and multiple sevoflurane exposures during pregnancy and offspring behavior in mice. Paediatr Anaesth. 2017 Jul;27(7):742-751. doi: 10.1111/pan.13139. Epub 2017 May 11. PMID 28497474
- [Result] Yeo ST, Holdcroft A, Yentis SM, Stewart A. Analgesia with sevoflurane during labour: i. Determination of the optimum concentration. Br J Anaesth. 2007 Jan;98(1):105-9. doi: 10.1093/bja/ael326. PMID 17158128
- [Result] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins--Obstetrics. Practice Bulletin No. 161: External Cephalic Version. Obstet Gynecol. 2016 Feb;127(2):e54-61. doi: 10.1097/AOG.0000000000001312. PMID 26942387
- [Result] Magro-Malosso ER, Saccone G, Di Tommaso M, Mele M, Berghella V. Neuraxial analgesia to increase the success rate of external cephalic version: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2016 Sep;215(3):276-86. doi: 10.1016/j.ajog.2016.04.036. Epub 2016 Apr 27. PMID 27131581
- [Result] Cluver C, Gyte GM, Sinclair M, Dowswell T, Hofmeyr GJ. Interventions for helping to turn term breech babies to head first presentation when using external cephalic version. Cochrane Database Syst Rev. 2015 Feb 9;2015(2):CD000184. doi: 10.1002/14651858.CD000184.pub4. PMID 25674710
- [Result] Goodman S. Anesthesia for nonobstetric surgery in the pregnant patient. Semin Perinatol. 2002 Apr;26(2):136-45. doi: 10.1053/sper.2002.32203. PMID 12005471
- [Result] Satomoto M, Satoh Y, Terui K, Miyao H, Takishima K, Ito M, Imaki J. Neonatal exposure to sevoflurane induces abnormal social behaviors and deficits in fear conditioning in mice. Anesthesiology. 2009 Mar;110(3):628-37. doi: 10.1097/ALN.0b013e3181974fa2. PMID 19212262
- [Result] Song R, Ling X, Peng M, Xue Z, Cang J, Fang F. Maternal Sevoflurane Exposure Causes Abnormal Development of Fetal Prefrontal Cortex and Induces Cognitive Dysfunction in Offspring. Stem Cells Int. 2017;2017:6158468. doi: 10.1155/2017/6158468. Epub 2017 Sep 25. PMID 29098009
- [Result] Zheng H, Dong Y, Xu Z, Crosby G, Culley DJ, Zhang Y, Xie Z. Sevoflurane anesthesia in pregnant mice induces neurotoxicity in fetal and offspring mice. Anesthesiology. 2013 Mar;118(3):516-26. doi: 10.1097/ALN.0b013e3182834d5d. PMID 23314109
- [Result] Fok WY, Chan LW, Leung TY, Lau TK. Maternal experience of pain during external cephalic version at term. Acta Obstet Gynecol Scand. 2005 Aug;84(8):748-51. doi: 10.1111/j.0001-6349.2005.00505.x. PMID 16026399
- [Result] Yildiz K, Dogru K, Dalgic H, Serin IS, Sezer Z, Madenoglu H, Boyaci A. Inhibitory effects of desflurane and sevoflurane on oxytocin-induced contractions of isolated pregnant human myometrium. Acta Anaesthesiol Scand. 2005 Oct;49(9):1355-9. doi: 10.1111/j.1399-6576.2005.00804.x. PMID 16146475
- [Result] Wang ZH, Yang Y, Xu GP. Remifentanil analgesia during external cephalic version for breech presentation in nulliparous women at term: A randomized controlled trial. Medicine (Baltimore). 2017 Mar;96(11):e6256. doi: 10.1097/MD.0000000000006256. PMID 28296735
- [Result] Munoz H, Guerra S, Perez-Vaquero P, Valero Martinez C, Aizpuru F, Lopez-Picado A. Remifentanil versus placebo for analgesia during external cephalic version: a randomised clinical trial. Int J Obstet Anesth. 2014 Feb;23(1):52-7. doi: 10.1016/j.ijoa.2013.07.006. Epub 2014 Jan 3. PMID 24388737
- [Result] Khaw KS, Lee SW, Ngan Kee WD, Law LW, Lau TK, Ng FF, Leung TY. Randomized trial of anaesthetic interventions in external cephalic version for breech presentation. Br J Anaesth. 2015 Jun;114(6):944-50. doi: 10.1093/bja/aev107. Epub 2015 May 10. PMID 25962611
- [Result] Weiniger CF, Ginosar Y, Elchalal U, Sela HY, Weissman C, Ezra Y. Randomized controlled trial of external cephalic version in term multiparae with or without spinal analgesia. Br J Anaesth. 2010 May;104(5):613-8. doi: 10.1093/bja/aeq053. Epub 2010 Mar 25. PMID 20338954
- [Result] Chalifoux LA, Bauchat JR, Higgins N, Toledo P, Peralta FM, Farrer J, Gerber SE, McCarthy RJ, Sullivan JT. Effect of Intrathecal Bupivacaine Dose on the Success of External Cephalic Version for Breech Presentation: A Prospective, Randomized, Blinded Clinical Trial. Anesthesiology. 2017 Oct;127(4):625-632. doi: 10.1097/ALN.0000000000001796. PMID 28723831